CLINICAL TRIAL: NCT06337721
Title: Preventing Alcohol Use Disorders and Alcohol-Related Harms in Pacific Islander Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AA030786 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Use Disorder; Alcohol; Harmful Use
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Will conduct a randomized controlled trial of the SPEAR intervention vs. control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPEAR (Experimental): This arm will consist of the SPEAR (Strategies for Pacific Empowerment and Alcohol Reduction) behavioral group intervention to reduce AUDs and alcohol-related harms in Pacific Islander young adults.
  Interventions: Behavioral: SPEAR (Strategies for Pacific Empowerment and Alcohol Reduction)
- Control (No Intervention): This control group arm will be compared to the SPEAR intervention.

INTERVENTIONS:
Behavioral: SPEAR (Strategies for Pacific Empowerment and Alcohol Reduction) — This behavioral group intervention will consist of multiple group sessions to reduce AUDs and alcohol-related harms in Pacific Islander young adults. It will infuse culturally resonant narratives, language, and elements into existing evidence-based strategies.
  Arms: SPEAR

SUMMARY:
This study will: (1) refine and finalize the SPEAR intervention manual for preventing alcohol use disorders (AUD) and associated harms for Pacific Islander young adults; and (2) test SPEAR for efficacy by conducting a pretest-posttest randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Pacific Islander young adults bear elevated risk for alcohol use disorders (AUD) and alcohol-related harms, yet lack effective interventions to reduce their risk. Grounded in the social development model, this study will: (1) refine and finalize the SPEAR intervention manual for preventing alcohol use disorders (AUD) and associated harms for Pacific Islander young adults from existing evidence-based AUD prevention strategies; then (2) test SPEAR for efficacy by conducting a pretest-posttest randomized controlled trial (RCT) with at-risk Pacific Islander young adults across multiple Pacific Islander communities in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Of full or part self-reported Pacific Islander heritage;
2. Fluent (oral and reading) in English
3. For young adult participants: 18 - 30 years of age
4. Current drinking (1+ drink in past 30 days)
5. High AUD risk (AUDIT-C score # 4 for men, # 3 for women)
6. Not currently in alcohol treatment (medication, therapeutic).

Exclusion Criteria:

1. Do not meet inclusion criteria
2. Are unwilling to participate
3. Fail to provide or retracts consent
4. Reside outside the target Pacific Islander communities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Heavy Episodic Drinking (HED) Days | Up to 30 weeks
  # of Days of HED out of past 30 days

SECONDARY OUTCOMES:
Alcohol Consumption | Up to 30 weeks
  7-day Alcohol Consumption

CONTACTS AND LOCATIONS:
Overall Officials: ANDREW SUBICA, Principal Investigator — UC Riverside
Locations (1):
- UC Riverside, Riverside, California, United States